**Study Title:** Effect of bisphosphonate use on surgical weight loss associated bone loss in older adults with morbid obesity (WEight loss with RISEdronate for bone health; **WE RISE**)

IRB00048310 NCT03411902 Date: 12/29/20

Principal Investigator, Co-investigator(s): Co-PIs: Kristen Beavers and Jamy Ard. Co-Is: Adolfo

Fernandez, Daniel Beavers, Ashley Weaver, and Laura Flores

## Statistical Analysis Plan

Baseline characteristics were summarized overall and by randomized treatment group as means and standard deviations (mean±SD) for continuous variables or counts and percentages [n (%)] for discrete variables. Treatment effects of risedronate versus placebo were estimated using a mixed linear model fit with treatment assignment, visit, and treatment by visit interaction, adjusted for baseline characteristics of each outcome and assuming an unstructured covariance. Groups were compared using contrast statements at six and 12 months, with change over six months being the primary comparison. All statistical analyses were performed using SAS v9.4 (SAS Institute, Cary, NC) with significance based on a Type I error rate of 0.05. Because the study was designed as a pilot to determine feasibility and gather evidence for future work, analyses were not adjusted for multiple outcomes, and findings are not considered confirmatory.